CLINICAL TRIAL: NCT07125898
Title: Decoding Central Defects in Dystrophinopathies From Diagnostic to Remediation
Acronym: DECODYS
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP241376
Record Dates: First submitted 2025-08-11; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Dystrophinopathies
Keywords: Cognitive deficits; Autism-spectrum disorders; Attention deficit hyperactivity Disorder
MeSH Terms: conditions — Cognition Disorders; Child Development Disorders, Pervasive; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: PHASE 1: DMD diagnosis confirmed by a genetic analysis
- Group 2: PHASE 2: DMD diagnosis confirmed whose neuropsychological data are eligible for remediation

SUMMARY:
The study aims to identify a genotype/phenotype correlation by analyzing more finely the neurodevelopmental disorders in DMD patients.

DETAILED DESCRIPTION:
We propose a unique longitudinal study in which DMD children aged 5-12 years old will first be engaged in a deep evaluation of a range of cognitive, behavioral, physiological and neural functions (identification of biomarkers based on ERG) and an eligible subgroup of patients will then enter a second study phase (last 2 years) aimed at developing targeted cognitive remediation strategies:

1. Deep evaluation with research of correlation between DMD patients' genotype and neurological/neuropsychological phenotype: - the nature and severity of the cognitive/executive/behavioral deficits, - the retinal/visual alterations, - functional brain imaging.
2. Targeted cognitive remediation strategies in the same patients, to alleviate the identified neuropsychological and behavioral disturbances. We will place a particular focus on the socio-cognitive and executive weaknesse.

ELIGIBILITY:
Inclusion Criteria:

* French citizenship, affiliated to the French Social Security,
* 5 to 12 years old,
* DMD diagnosis confirmed by a genetic analysis predicting breaking in the reading frame of the DMD gene with knowledge of the limits of the mutation,
* Follow-up in a French referral or a skills center belonging to Filnemus.

Exclusion Criteria:

* Severe intellectual deficiency with IQ < 55, and IQ < 70 for the deep neurocognitive evaluation (executive and socio-cognitive evaluation),
* Cataract except if operated (pseudophakic),
* High intraocular pressure,
* Cardiac dysfunction with left ventricular ejection fraction < 35%,
* Respiratory dysfunction with force vital capacity < 70%,
* Difficulties in fine motor skills with D3 MFM scale < 75%
* Treatment with methylphenidate: In case of hyperactive patients, the treatment will be transitorily interrupted the week before testing.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: DMD diagnosis confirmed by a genetic analysis
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Nature and severity of sensory and neuropsychological disturbances | 12 Months
  Specify the nature and severity of sensory and neuropsychological disturbances (cognitive, executive, emotional, behavioral and neuropsychiatric) according to the patient's genotype.

SECONDARY OUTCOMES:
Correlations between sensory and neuropsychological measures | 24 Months
  Analyze the correlations between sensory (retinal/visual) and neuropsychological measures, in order to determine if retinal defects represent a signature of neuropsychological impairment severity.
Correlation between neuropsychological and functional imaging parameters | 24 Months
  Analyze correlation between neuropsychological and functional imaging parameters.
Correlation between sensory and functional imaging parameters | 24 Months
  Analyze correlation between sensory and functional imaging parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle DESGUERRE, MD, PhD, Principal Investigator — Hôpital Universitaire Necker - Enfants Malades
Locations (1):
- Hôpital Necker Enfants Malades, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No